CLINICAL TRIAL: NCT05479565
Title: The Association of Reduced Arterial Stiffness and Highly Sensitive C-reactive Protein With Gestational Diabetes Mellitus.
Brief Title: Relationship of Reduced Arterial Stiffness and Hs-CRP With GDM.
Status: Completed | Type: Observational
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Ana Dugandžić Šimić, mr. sc. Ana Dugandžić Šimić, ob/gyn specialist, University of Mostar
Other Study IDs: Arterial stiffness, GDM
Record Dates: First submitted 2022-07-14; First posted 2022-07-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 50 pregnant women with patological OGTT: 50 pregnant women with patological OGTT ( glucose load test) and after delivery - 50 women with GDM in previous pregnancy.
  Interventions: Diagnostic Test: venous blood sample for determining the value of highly sensitive C-reactive C protein from serum
- 50 pregnant women with regular OGTT: 50 pregnant women with regular OGTT ( glucose load test) and after delivery - 50 women without GDM in previous pregnancy
  Interventions: Diagnostic Test: venous blood sample for determining the value of highly sensitive C-reactive C protein from serum

INTERVENTIONS:
Diagnostic Test: venous blood sample for determining the value of highly sensitive C-reactive C protein from serum — The non-invasive oscillometric device Arteriograph (TensioMedTM Kft, Budapest, Hungary) will be used to measure the arterial stiffness. In a quiet room at room temperature, the subjects will lie relaxed for 15 minutes before the start of the measurement. After that, the distance between the jugulum and the symphysis, which represents the approximate length of the aorta, will be measured with a gynecological compass, and the resulting value will be entered into the device.
  Other Names: measuring the arterial stiffness

SUMMARY:
Research hypotheses

1. The arterial stiffness in pregnant women with gestational diabetes is reduced compared to healthy pregnant women.
2. The values of highly sensitive CRP in pregnant women with gestational diabetes are higher compared to healthy pregnant women.
3. The arterial stiffness in test subjects with previous gestational diabetes was reduced compared to test subjects with a previously normal OGTT during pregnancy.
4. The values of highly sensitive CRP in subjects with previous gestational diabetes are higher compared to subjects with previously normal OGTT during pregnancy.

DETAILED DESCRIPTION:
Gestational diabetes is a growing problem at the global level, and it brings with it numerous perinatal and maternal complications. In addition, it is associated with a higher risk of developing type 2 diabetes and cardiovascular disease later in life. However, the mechanisms by which this happens have not been fully elucidated, which is why the possibilities of prevention are limited. Insulin resistance is recognized as a cause of GDM and associated with a decrease in arterial elasticity due to its pro-inflammatory pathogenesis, which is manifested by an increase in pro-inflammatory biomarkers, such as hs CRP. However, the application of these findings has not yet taken root in practice.

It is necessary to find reliable methods of screening pregnant women with GDM who have an increased risk of developing complications both during pregnancy and later in life.

Reduced arterial elasticity is recognized as a predictor of cardiovascular diseases, and its measurement is recommended to be introduced into clinical practice. On the other hand, measuring hsCRP is simple and available, but its practical application is still questionable and additional research is needed. Several studies have attempted to link GDM with reduced arterial elasticity and/or increased hs CRP, but the conclusions are contradictory, probably due to the small number of subjects. On the other hand, I did not find studies that measured the mentioned parameters just after delivery for the purpose of predicting cardiovascular risk (80-82 ref from MR).

This research will try to prove the association of GDM with reduced arterial stiffness and elevated hsCRP values. The results will attempt to justify the introduction into clinical practice of measuring arterial elasticity and hsCRP in order to find pregnant women at risk of developing complications during and after pregnancy.

Research objectives

Main goals:

* To compare the arterial stiffness in pregnant women with gestational diabetes and healthy pregnant women.
* To compare the values of highly sensitive CRP in pregnant women with gestational diabetes and healthy pregnant women
* To determine whether the occurrence of cardiovascular diseases during pregnancy can be predicted by measuring the arterial stiffness and hs CRP in healthy pregnant women and pregnant women with GDM

Secondary objectives:

* To compare the occurrence of pregnancy complications and perinatal outcome in pregnant women with gestational diabetes and healthy pregnant women.
* To compare the srterial stiffness and the values of highly sensitive CRP in two groups of subjects 2-6 months after pregnancy.

The purpose of the research

Measurement of arterial stiffness and high-sensitivity CRP values could, based on the results of this study, be introduced into clinical practice as predictors of GDM-related complications in pregnancy and later in life.

Research hypotheses

1. The arterial stiffness in pregnant women with gestational diabetes is reduced compared to healthy pregnant women.
2. The values of highly sensitive CRP in pregnant women with gestational diabetes are higher compared to healthy pregnant women.
3. The arterial stiffness in test subjects with previous gestational diabetes was reduced compared to test subjects with a previously normal OGTT during pregnancy.
4. The values of highly sensitive CRP in subjects with previous gestational diabetes are higher compared to subjects with previously normal OGTT during pregnancy.

Respondents:

1. 100 pregnant women from the 28th to the 40th week of pregnancy (in the third trimester), who, as part of regular perinatal care, took the oral glucose tolerance test (OGTT), divided into two groups:

   * 50 pregnant women with pathological findings of OGTT i
   * 50 pregnant women with regular OGTT.

   The diagnosis of gestational diabetes will be made on the basis of the pathological findings of the OGTT, according to WHO criteria from 2013: the OGTT will be performed with 75 g of glucose, and it is sufficient that only one of the stated concentrations of glucose taken from the mother's venous blood plasma is equal to or higher from borderline:
   * fasting glycemia ≥ 5.1 mmol/l,
   * glycemia after 1h ≥ 10 mmol/l,
   * glycemia after 2h ≥ 8.5mmol/l.

   At the same time, the glycemic values must not meet the criteria for manifest diabetes:
   * fasting glycemia ≥ 7.0 mmol/l,
   * glycemia after 2 h ≥ 11.1 mmol/l,
   * glycemia at any time ≥ 11.1 mmol/l with the presence of diabetes symptoms.

   Criteria for the inclusion of test subjects:
   * age between 18 and 35 years
   * previously healthy women
   * previously normal course of pregnancy
   * singleton pregnancies
   * non-smokers

   Exclusion criteria:
   * pregestational diabetes
   * gestational diabetes and/or hypertensive disorders in pregnancy in previous pregnancies
   * hypertensive disorders during pregnancy at the time of examination
   * chronic diseases
   * pregnant women whose partner previously had a partner with preeclampsia.
2. Two to six months after delivery of the same test subjects, divided into the same two groups: 50 test subjects with previous normal OGTT during pregnancy and 50 test subjects with previous gestational diabetes.

The test subjects will have a venous blood sample taken to determine the value of highly sensitive C-reactive C protein from the serum and measure the arterial stiffness.

The non-invasive oscillometric device Arteriograph (TensioMedTM Kft, Budapest, Hungary) will be used to measure the arterial stiffness.

The indicators of arterial stiffnesses, which will be used in the analysis, will be:

* pulse wave speed,
* central systolic pressure,
* peripheral and central values of the augmentation index,
* peripheral and central pulse pressure values.

Pregnant women will then be monitored until delivery, in order to determine whether they will develop the following pregnancy complications:

* hypertensive disorders (gestational hypertension, preeclampsia, eclampsia)
* induction of labor (iatrogenic labor induction)
* operative completion of childbirth (caesarean section or vacuum extraction)

Also, it will be determined what the perinatal outcome of the newborn will be, i.e. whether there will be:

* macrosomia (newborn weight above 4000 g),
* a newborn large for gestational age, a newborn weighing more than the 90th percentile for gestational age.
* trauma during childbirth (shoulder dystocia, clavicle fracture, brachial plexus injuries),
* metabolic disorders of the newborn (hypoglycemia, hypomagnesemia, hypocalcemia, hyperviscosity syndrome, occurrence of neonatal jaundice),
* stay in the Neonatal Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* previously healthy women
* previously normal course of pregnancy
* singleton pregnancies
* non-smokers

Exclusion Criteria:

* pregestational diabetes
* gestational diabetes and/or hypertensive disorders in pregnancy in previous pregnancies
* hypertensive disorders during pregnancy at the time of examination
* chronic diseases
* pregnant women whose partner previously had a partner with preeclampsia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: * age between 18 and 35 years
  * previously healthy women
  * previously normal course of pregnancy
  * singleton pregnancies
  * non-smokers
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The arterial stiffness in pregnant women with gestational diabetes is reduced compared to healthy pregnant women. | between 28 and 40 weeks of gestation
  The non-invasive oscillometric device Arteriograph will be used to measure the arterial stiffness.The examiners will use a gynecological divider to measure the distance between the jugulum and the symphysis, which represents the approximate length of the aorta, and the obtained value will be entered into the device
The values of highly sensitive CRP in pregnant women with gestational diabetes are higher compared to healthy pregnant women. | between 28 and 40 weeks of gestation
  The test subjects will have a venous blood sample taken to determine the value of highly sensitive C-reactive C protein from the serum.

CONTACTS AND LOCATIONS:
Overall Officials: Vajdana Tomić, prof.dr.sc., Study Chair — Faculty of Health Studies, Mostar
Locations (1):
- University of Mostar, Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 Years folowing article publication.
Access Criteria: Investigators whose proposed use the Data has been approved by an Independent review committee identified for this purpose.